CLINICAL TRIAL: NCT00209053
Title: A Prospective, Randomized Comparison of Graft Patency and Clinical Outcomes After Coronary Bypass Surgery Performed With and Without the Use of Cardiopulmonary Bypass:Longitudinal Follow-Up
Brief Title: SMART Trial Longitudinal Follow-Up:Off-Pump Versus On-Pump Coronary Artery Bypass Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: Medtronic (Industry); Boston Scientific Corporation (Industry)
Responsible Party: Principal Investigator, John Puskas, MD, Professor, Emory University
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: 0517-1999
Record Dates: First submitted 2005-09-14; First posted 2005-09-21 (Estimated); Last update posted 2013-10-16 (Estimated); Status verified 2013-10

CONDITIONS: Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease | interventions — Coronary Artery Bypass

ARMS (2):
- Off Pump CABG (Experimental): CABG without cardiopulmonary bypass.
  Interventions: Procedure: Coronary Artery Bypass
- On-Pump CABG (Active Comparator): CABG with cardiopulmonary bypass.
  Interventions: Procedure: Coronary Artery Bypass

INTERVENTIONS:
Procedure: Coronary Artery Bypass

SUMMARY:
The purpose of this study is to determine completeness of revascularization, graft patency, clinical outcomes, health-related quality of life and costs in 200 initial trial participants at > 5 years post surgery who had heart bypass surgery with heart-lung bypass (on-pump) or without heart-lung bypass (off-pump). The hypothesis is that the patency of coronary artery bypass grafts of off-pump surgery are no less durable than grafts from conventional on-pump surgery.

DETAILED DESCRIPTION:
The Surgical Management of Arterial Revascularization Therapies (SMART) trial is a randomized, controlled, double blinded trial designed to compare completeness of revascularization, graft patency, clinical outcomes, health-related quality of life and costs in 200 unselected patients referred for elective, isolated coronary bypass surgery and randomized to have coronary artery bypass performed with or without cardiopulmonary bypass. These patients were enrolled between March 2000 to August 2001.

The primary objective of this study is to test the hypothesis that the patency of coronary artery bypass grafts constructed during off-pump coronary artery bypass (OPCAB)are no less durable than the patency of those constructed during conventional CABG with cardiopulmonary bypass (CABG/CPB)after > 5 years of follow-up (non-inferiority hypothesis).

The secondary objectives are to determine whether there are differences between these randomized groups in the following outcomes measures at > 5 years:

1. Neurocognitive Function
2. Stroke/cerebral injury
3. Health-related quality of life
4. Myocardial perfusion and ischemia
5. Major Adverse Cardiac Events (MACE)
6. Cardiac Functional Status
7. Incidence and severity of angina
8. All cause mortality and cardiovascular mortality
9. Cost of hospital re-admissions since 1 year follow-up

ELIGIBILITY:
Inclusion Criteria:

* Referred for primary or re-operative elective coronary artery bypass graft (CABG) with coronary targets suitable for off-pump bypass graft and currently enrolled in Phase 1 of SMART Trial

Exclusion Criteria:

* Emergent CABG
* Required pre-operative intra-aortic balloon pump (IABP)
* Cardiogenic shock
* Evolving acute myocardial infarction
* Coronary artery targets unsuitable for off-pump bypass surgery
* Inability or unwillingness to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 87 (Actual)
Dates: Start 2007-01; Primary Completion 2009-03 (Actual); Study Completion 2009-03 (Actual)

PRIMARY OUTCOMES:
after > 5 years, graft patency determined by non-invasive dual 64 slice multi-detector computed tomographic coronary angiography and cardiac positron emission tomography. | 8 year follow-up

SECONDARY OUTCOMES:
Secondary outcomes will be measured by; a battery of neuropsychological tests, MRI, NIH stroke scale, questionnaires, cardiac PET scanning, NYHA and CCS classifications and Medicare DRG's. | 8 year follow-up

CONTACTS AND LOCATIONS:
Overall Officials: John D Puskas, M.D., Principal Investigator — Emory University
Locations (1):
- Emory Healthcare/EmoryUniversity, Atlanta, Georgia, United States